CLINICAL TRIAL: NCT01406717
Title: Safety and Efficacy of SPIL1033 in Subjects With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sun Pharmaceutical Industries Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CLR_10_33
Record Dates: First submitted 2011-07-28; First posted 2011-08-01 (Estimated); Results first posted 2019-11-01 (Actual); Last update posted 2020-08-11 (Actual); Status verified 2020-07

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: SPIL1033; type 2 diabetes mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- SPIL1033 (Experimental)
  Interventions: Drug: SPIL1033
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SPIL1033 — 5 mcg twice daily for the first 4 weeks and 10 mcg twice daily for the remaining 20 weeks. To be self-administered twice daily.
  Arms: SPIL1033
Drug: Placebo — 5 mcg twice daily for the first 4 weeks and 10 mcg twice daily for the remaining 20 weeks. To be self-administered twice daily.
  Arms: Placebo

SUMMARY:
SPIL1033 resembles a gut hormone, which increases the insulin secretion, thus helps in reducing blood glucose levels. The purpose of study is to establish safety and efficacy of SPIL1033

DETAILED DESCRIPTION:
SPIL1033 is subcutaneous injection is indicated as adjunctive therapy to improve glycemic control in patients with type 2 diabetes mellitus.

In this study, efficacy and safety of SPIL1033 will be evaluated. Subjects will receive SPIL1033 or placebo, 5 mcg twice daily for the first 4 weeks and 10 mcg twice daily for the remaining 20 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects 20 years of age and older.
* Established clinical diagnosis of type 2 diabetes mellitus treated with diet and exercise or anti-diabetic agents as monotherapy or combination therapy.
* Weight stable: their weight should not have varied more than 10% of screening visit weight, within 6 months prior to screening visit.
* Women of child bearing potential practicing an acceptable method of birth control as judged by the investigator(s); with a negative urine pregnancy test.
* Willing to participate and give written informed consent.

Exclusion Criteria:

* Previous exposure to exenatide (anti-exenatide antibodies at screening) or a glucagon-like peptide (GLP-1) analogue.
* Used drugs for weight loss (for example, orlistat, sibutramine, phenylpropanolamine, rimonabant, or similar over-the-counter medications) within 3 months of screening.
* Received treatment within the last 30 days with a drug that has not received regulatory approval for any indication at the time of trial entry.
* Severe renal impairment (creatinine clearance <30 ml/min) or end stage renal disease.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Actual)
Dates: Start 2013-03-01; Primary Completion 2015-11-04 (Actual); Study Completion 2015-11-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (34):
- India (34):
  - SPIL Site 22, Hyderabad, Andhra Pradesh
  - SPIL Site 25, Hyderabad, Andhra Pradesh
  - SPIL Site 26, Hyderabad, Andhra Pradesh
  - SPIL Site 23, Visakhapatnam, Andhra Pradesh
  - SPIL Site 1, Ahmedabad, Gujarat
  - SPIL Site 2, Ahmedabad, Gujarat
  - SPIL Site 3, Ahmedabad, Gujarat
  - SPIL Site 5, Rajkot, Gujarat
  - SPIL Site 6, Surat, Gujarat
  - SPIL Site 7, Surat, Gujarat
  - SPIL Site 8, Surat, Gujarat
  - SPIL Site 9, Surat, Gujarat
  - SPIL Site 10, Vadodara, Gujarat
  - SPIL Site 19, Bangalore, Karnataka
  - SPIL Site 30, Bangalore, Karnataka
  - SPIL Site 31, Bangalore, Karnataka
  - SPIL Site 33, Bangalore, Karnataka
  - SPIL Site 29, Manipal, Karnataka
  - SPIL Site 35, Indore, Madhya Pradesh
  - SPIL Site 21, Nagpur, Maharashtra
  - SPIL Site 24, Nagpur, Maharashtra
  - SPIL Site 32, Nashik, Maharashtra
  - SPIL Site 11, Pune, Maharashtra
  - SPIL Site 12, Pune, Maharashtra
  - SPIL Site 13, Bhubaneshwar, Orrissa
  - SPIL Site 14, Jaipur, Rajasthan
  - SPIL Site 15, Jaipur, Rajasthan
  - SPIL Site 16, Chennai, Tamil Nadu
  - SPIL Site 17, Coimbatore, Tamil Nadu
  - SPIL Site 20, Coimbatore, Tamil Nadu
  - SPIL Site 18, Madurai, Tamil Nadu
  - SPIL Site 34, Vellore, Tamil Nadu
  - SPIL Site 27, Lucknow, Uttar Pradesh
  - SPIL Site 28, Lucknow, Uttar Pradesh

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | SPIL1033 | Placebo
Started | 180 | 180
Completed | 137 | 149
Not Completed | 43 | 31
Not completed — Subject non-compliance | 4 | 3
Not completed — Protocol Violation | 5 | 1
Not completed — Lost to Follow-up | 14 | 8
Not completed — Withdrawal by Subject | 19 | 15
Not completed — Adverse Event | 1 | 2
Not completed — Lack of Efficacy | 0 | 1
Not completed — Non-completion of visit activity | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- SPIL1033: SPIL1033: 5 mcg twice daily for the first 4 weeks and 10 mcg twice daily for the remaining 20 weeks. To be self-administered twice daily.
  168 are the number of subjects in mITT population
- Placebo: Placebo: 5 mcg twice daily for the first 4 weeks and 10 mcg twice daily for the remaining 20 weeks. To be self-administered twice daily.
  170 are the number of subjects in mTT population.
- Total: Total of all reporting groups
Arm/Group | SPIL1033 | Placebo | Total
Number analyzed (Participants) | 168 | 170 | 338
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.9 (9.26) | 51.9 (9.56) | 52.4 (9.41)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 83 | 86 | 169
  Male | 85 | 84 | 169
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 168 | 170 | 338
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to End of Study in Hemoglobin A1c (HbA1c)
Time Frame: 24 weeks
Population: Intent-to-treat
Measure: Least Squares Mean (Standard Error); unit: percentage of hemoglobin A1c (HbA1c)
Groups:
- SPIL1033: SPIL1033: 5 mcg twice daily for the first 4 weeks and 10 mcg twice daily for the remaining 20 weeks. To be self-administered twice daily. The number of subjects in evaluable population for efficacy (EPE) population are 112.
- Placebo: Placebo: 5 mcg twice daily for the first 4 weeks and 10 mcg twice daily for the remaining 20 weeks. To be self-administered twice daily. The number of subjects in evaluable population for efficacy (EPE) population are 94.
Arm/Group | SPIL1033 | Placebo
Number analyzed (Participants) | 112 | 94
percentage of hemoglobin A1c (HbA1c) | -0.227 (0.243) | -0.227 (0.254)
Statistical Analysis 1: Comparison: SPIL1033 vs Placebo; Test type: Other; ANCOVA = 0.0002, 95% CI 2-sided [-0.31377 to 0.31418]

2. Primary Outcome: Change From Baseline to End of Study in Fasting Plasma Glucose (FPG)
Time Frame: 24 weeks
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Groups:
- SPIL1033: SPIL1033, Placebo: 5 mcg twice daily for the first 4 weeks and 10 mcg twice daily for the remaining 20 weeks. To be self-administered twice daily. he number of subjects in the population for the analysis of FPG are 110.
- Placebo: SPIL1033, Placebo: 5 mcg twice daily for the first 4 weeks and 10 mcg twice daily for the remaining 20 weeks. To be self-administered twice daily. he number of subjects in the population for the analysis of FPG are 94.
Arm/Group | SPIL1033 | Placebo
Number analyzed (Participants) | 110 | 94
mg/dL | 0.48 (9.78) | -5.42 (10.21)
Statistical Analysis 1: Comparison: SPIL1033 vs Placebo; Test type: Other; ANCOVA = 5.898, 95% CI 2-sided [-6.7565 to 18.5535]

3. Primary Outcome: Count and Percentage of Subjects Positive for Anti-exenatide Antibodies
Time Frame: 24 weeks
Population: modified intent to treat population
Measure: Count of Participants; unit: Participants
Groups:
- SPIL1033: SPIL1033: 5 mcg twice daily for the first 4 weeks and 10 mcg twice daily for the remaining 20 weeks. To be self-administered twice daily. The number of subjects in the evaluated anti-exenatide antibodies are 133.
- Placebo: Placebo: 5 mcg twice daily for the first 4 weeks and 10 mcg twice daily for the remaining 20 weeks. To be self-administered twice daily. The number of subjects in evaluated anti-exenatide antibodies population are 143.
Arm/Group | SPIL1033 | Placebo
Number analyzed (Participants) | 133 | 143
Participants | 59 | 2
Statistical Analysis 1: Comparison: SPIL1033 vs Placebo; Test type: Other; p < 0.0001, Mantel Haenszel

4. Primary Outcome: Count and Percentage of Subjects With Potentially Immune-related Treatment-emergent Adverse Events (TEAEs)
Time Frame: 24 weeks
Population: Evaluable population for safety: subjects who were randomized and received at least one dose of a trial medication
Measure: Count of Participants; unit: Participants
Groups:
- SPIL1033: SPIL1033: 5 mcg twice daily for the first 4 weeks and 10 mcg twice daily for the remaining 20 weeks. To be self-administered twice daily. The number of subjects in the safety population are 179.
- Placebo: Placebo: 5 mcg twice daily for the first 4 weeks and 10 mcg twice daily for the remaining 20 weeks. To be self-administered twice daily. The number of subjects in the safety population are 178.
Arm/Group | SPIL1033 | Placebo
Number analyzed (Participants) | 179 | 178
Participants | 3 | 3

5. Secondary Outcome: Change From Baseline in 2hour Postprandial Glucose (2-h PPG)
Time Frame: 24 weeks
Population: The evaluable population: all mITT subjects who received at least 80% of study medication over 24 weeks and completed treatment through week 24. (modified Intent-to-treat population: .subjects who were randomized and received at least one dose of the trial medication after visit 2 (baseline) and had at least one post-baseline visit.
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | SPIL1033 | Placebo
Number analyzed (Participants) | 139 | 148
mg/dl | -21.20 (14.50) | -16.83 (14.49)
Statistical Analysis 1: Comparison: SPIL1033 vs Placebo; Test type: Other; p = 0.6318, ANCOVA

6. Secondary Outcome: Change From Baseline in Triglycerides
Time Frame: 24 weeks
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: mg/dl
Arm/Group | SPIL1033 | Placebo
Number analyzed (Participants) | 143 | 150
mg/dl | 1.27 (16.53) | 8.39 (16.53)
Statistical Analysis 1: Comparison: SPIL1033 vs Placebo; Test type: Other; p = 0.4887, ANOVA

7. Secondary Outcome: Change From Baseline in Low Density Lipoproteins
Time Frame: 24 weeks
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | SPIL1033 | Placebo
Number analyzed (Participants) | 143 | 150
mg/dL | -3.18 (6.12) | 0.15 (6.12)
Statistical Analysis 1: Comparison: SPIL1033 vs Placebo; Test type: Other; p = 0.3813, ANOVA

8. Secondary Outcome: Change From Baseline in High Density Lipoproteins
Time Frame: 24 weeks
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | SPIL1033 | Placebo
Number analyzed (Participants) | 143 | 149
mg/dL | 0.64 (2.16) | 0.62 (2.16)
Statistical Analysis 1: Comparison: SPIL1033 vs Placebo; Test type: Other; p = 0.9900, ANOVA

9. Secondary Outcome: Change in Body Weight
Time Frame: 24 weeks
Measure: Least Squares Mean (Standard Error); unit: kilograms
Arm/Group | SPIL1033 | Placebo
Number analyzed (Participants) | 143 | 153
kilograms | -1.708 (0.468) | -0.792 (0.467)
Statistical Analysis 1: Comparison: SPIL1033 vs Placebo; Test type: Other; p = 0.0017, ANOVA

10. Secondary Outcome: Subjects Achieving Hemoglobin A1c (HbA1c) < 7%
Time Frame: 24 weeks
Population: Evaluable Population for Efficacy
Measure: Count of Participants; unit: Participants
Groups:
- SPIL1033: SPIL1033: 5 mcg twice daily for the first 4 weeks and 10 mcg twice daily for the remaining 20 weeks. To be self-administered twice daily. The number of subjects in the population for the analysis of HbA1c are 112.
- Placebo: Placebo: 5 mcg twice daily for the first 4 weeks and 10 mcg twice daily for the remaining 20 weeks. To be self-administered twice daily. he number of subjects in the population for the analysis of HbA1c are 94.
Arm/Group | SPIL1033 | Placebo
Number analyzed (Participants) | 112 | 94
Participants | 26 | 20
Statistical Analysis 1: Comparison: SPIL1033 vs Placebo; Test type: Other; p = 0.6098, Mantel Haenszel

11. Secondary Outcome: Change From Baseline in Very Low Density Lipoproteins
Time Frame: 24 weeks
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | SPIL1033 | Placebo
Number analyzed (Participants) | 141 | 149
mg/dL | 0.88 (3.13) | 1.55 (3.13)
Statistical Analysis 1: Comparison: SPIL1033 vs Placebo; Test type: Other; p = 0.7324, ANOVA

12. Secondary Outcome: Change From Baseline in Total Cholesterol
Time Frame: 24 weeks
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | SPIL1033 | Placebo
Number analyzed (Participants) | 168 | 170
mg/dL | -4.89 (7.40) | -0.11 (7.40)
Statistical Analysis 1: Comparison: SPIL1033 vs Placebo; Test type: Other; p = 0.2984, ANOVA

ADVERSE EVENTS:
Arm/Group | SPIL1033 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/180 | 0/180
Serious Adverse Events (participants affected / at risk) | 6/180 | 1/180
Other Adverse Events (participants affected / at risk) | 126/180 | 115/180
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SPIL1033 (N=180) | Placebo (N=180)
Abscess limb (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0
Infected dermal cyst (Infections and infestations) | 1 | 0
Viral infection (Infections and infestations) | 1 | 0
joint injury (Injury, poisoning and procedural complications) | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0
Road traffic accident (Infections and infestations) | 1 | 0
Upper limb fracture (Infections and infestations) | 1 | 0
Hemiparesis (Nervous system disorders) | 0 | 1
Lumbar radiculopathy (Nervous system disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0
Gastroenteritis (Gastrointestinal disorders) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | SPIL1033 (N=180) | Placebo (N=180)
Hyperglycemia (Metabolism and nutrition disorders) | 52 | 59
Hypoglycaemia (Metabolism and nutrition disorders) | 17 | 11
Dyslipidaemia (Metabolism and nutrition disorders) | 19 | 13
Decreased appetite (Metabolism and nutrition disorders) | 11 | 2
Nausea (Gastrointestinal disorders) | 26 | 9
Diarrhoea (Gastrointestinal disorders) | 5 | 9
Vomiting (Gastrointestinal disorders) | 10 | 3
Headache (Nervous system disorders) | 13 | 8
Dizziness (Nervous system disorders) | 8 | 6
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 | 3
Back Pain (Musculoskeletal and connective tissue disorders) | 3 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other